CLINICAL TRIAL: NCT05473559
Title: Comparison Between i Pack Block and Post Tibial Nerve Block
Brief Title: Comparison Between the Effect of Infiltration Between the Popliteal Artery and Capsule of the Knee Block Versus Selective Tibial Nerve Block for Postoperative Analgesia in Patient Undergoing Total Knee Arthroplasty. A Prospective Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Abogabal, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 35151/12/21
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2021-12

CONDITIONS: Postoperative Analgesia

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adductor canal block with Ipack block (Active Comparator)
  Interventions: Procedure: Adductor canal block with Ipack block or selective tibial nerve block
- Adductor canal block with selective tibial nerve block (Active Comparator)
  Interventions: Procedure: Adductor canal block with Ipack block or selective tibial nerve block

INTERVENTIONS:
Procedure: Adductor canal block with Ipack block or selective tibial nerve block — Ultrasound guided

SUMMARY:
Comparison Between the Effect of Infiltration Between the Popliteal Artery and Capsule of the Knee Block Versus Selective Tibial Nerve Block for Postoperative Analgesia in Patient Undergoing Total Knee Arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis scheduled for a primary either partial or total knee arthroplasty • Patients aged 40-80 years with a body mass index of 18-36 kg/ m2 and an American Society of Anesthesiologists functional status of I-III Planned use of regional anesthesia

Exclusion Criteria:

* • Patients younger than 40 years old and older than 80years.

  * Hepatic or renal insufficiency.
  * Patients undergoing general anesthesia.
  * Allergy or intolerance to one of the study medications.
  * BMI > 36
  * Diabetes
  * ASA of IV
  * Chronic opioid use (taking opioids for longer than 3 months, or daily oral morphine equivalent of >5mg/day for one month)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours post operative
  24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Abogabal, MD, Principal Investigator — Tanta University; Wafaa Abdelwahed, MD, Principal Investigator — Tanta University; Wafaa Abdelsalam, MD, Principal Investigator — Kafr Elsheikh university; Shaimaa Zahra, Principal Investigator — Tanta University
Locations (1):
- Tanta university, Tanta, Egypt